CLINICAL TRIAL: NCT05466890
Title: Phase 2a, Double-Blind, Randomized Adaptive Design, Placebo-Controlled, Parallel Group Study to Evaluate the Safety, Tolerability, Efficacy, PK and Biomarkers with Oral Colon Delivery PL8177 in Adult Subjects with Active Ulcerative Colitis
Brief Title: Phase 2a to Evaluate PL-8177 in Subjects with Active Ulcerative Colitis (UC)
Acronym: PL8177-205
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Palatin Technologies, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PL8177-205
Record Dates: First submitted 2022-05-25; First posted 2022-07-20 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Ulcerative Colitis; Ulcerative Colitis Acute; Ulcerative; Ulcerative Colitis Flare
Keywords: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative; Ulcer

STUDY DESIGN:
Intervention Model Description: A non-stratified permuted block randomization scheme will be used to randomize the patients in a 3:1 ratio (PL8177: placebo).
Who Masked: Participant, Care Provider, Investigator
Masking Description: All trial participants, investigator sites, and Sponsor are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PL8177 (Experimental): PL8177 will be given orally and daily from baseline until end of study.
  Interventions: Drug: PL8177
- Placebo (Placebo Comparator): Approximately 1/4 of randomized patients will receive matching placebo as means of comparison to active treatment PL8177.
  Interventions: Drug: PL8177 Placebo

INTERVENTIONS:
Drug: PL8177 Placebo — Approximately 1/4 of randomized patients will receive matching placebo as means of comparison to active treatment PL8177.
  Other Names: Placebo
  Arms: Placebo
Drug: PL8177 — Approximately 3/4 of randomized patients will receive active PL8177.
  Other Names: Active study medication
  Arms: PL8177

SUMMARY:
The purpose of this study is to compare PL8177 (a melanocortin receptor agonist) to placebo (in a 3:1 ratio-meaning that for every 3 people that get the active drug, one will receive placebo). The study treatment will be for 8 weeks. The study will measure safety and the body's ability to handle PL8177 and look at the improvement and healing of the intestine after 8 weeks of treatment. The study will include adult males and nonpregnant, nonlactating females with acute Ulcerative Colitis (UC).

DETAILED DESCRIPTION:
This study will have potential subjects participating for approximately 4 months: Subjects will be screened to assess their eligibility within 28 days prior to the first dose administration; Day 1 will be eligibility confirmation and in-clinic dosing; additional visits to occur at Weeks 2, 4, 8 and 12. Routine laboratory tests, vital signs and ECG will be measured as well as blood, stool and tissue samples obtained for biomarker and PK studies. Endoscopy is required at screening visit and week 8 visit. Patients will also be given an electronic diary to enter on a daily basis for the duration of their participation. Additional patient questionnaires will be done at clinic visits. Optional genomics testing will also be completed for this study to help look at genes and their effect on inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 to ≤75 years of age at Screening.
* Has a history of UC diagnosis prior to screening; confirmed by endoscopic and histologic evidence in the subject chart. If the historical evidence is not available, then endoscopic and histologic evidence can be confirmed during the screening period.

Note: If no complete colonoscopy (adequate in quality to assess for dysplasia and colorectal polyps) has been performed and documented (with reports) within the past 1 year as recommended by local and national guidelines depending on Colorectal cancer risk factors in the specified subject, a full colonoscopy should be performed at screening. If such results are available within one year, a flexible sigmoidoscopy with examination up to the splenic flexure will be used for screening.

* Has active UC defined as a MES ≥2 during screening sigmoidoscopy.
* Has evidence of endoscopic disease extending to at least 5 cm proximal to the anal verge.
* If currently receiving 5-ASA, the duration and dose prior to the screening endoscopy must be as specified below, and a stable dose must be maintained throughout the double-blind trial: 5-aminosalicylates (5-ASA) (e.g., mesalamine, sulfasalazine, olsalazine, balsalazide) for ≥4 weeks with the dose stable for ≥3 weeks prior to the screening endoscopy.
* If recently has received any of the following treatments, they must have discontinued as specified below:

  * If 5-ASA has been recently discontinued, it must have been stopped for ≥3 weeks prior to the screening endoscopy.
  * If a thiopurine has recently been discontinued, it must have been stopped for ≥4 weeks prior to the screening endoscopy.
  * Oral corticosteroids must have been stopped for ≥4 weeks prior to the screening endoscopy.
* Women of childbearing potential must have a negative serum pregnancy test at screening and a negative urine pregnancy test at Day 1 prior to first dose of study drug.
* Male and female subjects of childbearing potential must agree to use 1 highly effective form of birth control during study participation and for 30 days after the last dose of study drug, unless the subject or his/her partner is surgically sterilized, or the subject agrees to abstain from sexual intercourse.
* Highly effective methods of birth control in this study include intrauterine device, hormonal contraceptives (oral, patch, long acting injectable, implant). Note: Oral hormonal contraceptives should be combined estrogen and progesterone. If a progesterone-only oral contraceptive is used, then a second method of birth control should be used as well.
* Postmenopausal is defined as lack of menses for ≥12 months prior to screening, confirmed by serum FSH >25 IU at Screening.
* Has provided informed consent prior to initiation of any study specific activities/procedures.
* Understands and is willing and able to comply with study requirements, including the schedule of events and follow-up visits.

Exclusion Criteria:

Subjects will be excluded from the study if they meet any of the following criteria at the Screening visit unless otherwise stated:

* Any condition, physical finding, laboratory or ECG abnormality, which, in the opinion of the Investigator, poses a safety risk, will prevent the subject from completing the study, will interfere with the interpretation of the study results, or might cause the study to be detrimental to the subject.
* Has fulminant colitis, toxic megacolon, microscopic colitis, history of colitis-associated colonic dysplasia, active peptic ulcer disease, cervical dysplasia, or primary sclerosing cholangitis.
* History of Crohn's disease or indeterminate colitis, or the presence or history of a fistula consistent with Crohn's disease.
* Presence of ileostomy or colostomy, or history of prior colon resection.
* Presence of adenomatous colonic polyps that have not been removed.
* Stools positive for C. difficile, enteric pathogens (Salmonella, Shigella, Campylobacter), or ova and parasites within 28 days of screening. Screen failures due to positive C. difficile or other enteric infection can be re-screened after appropriate treatment.
* History of mitochondrial disorder.
* History of primary or secondary immunodeficiency.
* History of cancer within the 5 years prior to screening including solid tumors and hematological malignancies (exception: no approval needed for basal cell and in situ squamous cell carcinomas of the skin that have been adequately treated with no re-occurrence for at least 1 year prior to screening).

History of one or more clinically relevant neurologic, psychologic, ophthalmologic, pulmonary, cardiovascular, gastrointestinal (other than the UC), hepatic, renal, endocrine, or other major systemic disease of moderate (or worse) severity, making implementation of the protocol or interpretation of the study difficult. Examples of (but not limited to) conditions to be excluded, are the following:

* Uncontrolled hypertension, with systolic blood pressure (SBP) ≥160 mmHg, diastolic blood pressure (DBP) ≥90 mmHg.
* Uncontrolled hyperlipidemia (even if therapy is ongoing, LDL>200 mg/dl or triglycerides >500 mg/dL).
* Known uncontrolled hyperthyroidism or hypothyroidism.
* Impaired hepatic function (Aspartate aminotransferase [AST] or Alanine aminotransferase [ALT] values >2.0 times the upper limit of the reference range and/or serum bilirubin >1.5 times the upper limit of the reference range at the screening visit).
* Cardiac or pulmonary disease, such as unstable angina or myocardial infarction within the past 12 months, congestive heart failure (CHF) Grade 2, 3, or 4 according to New York Heart Association criteria, valvular heart disease, cardiac arrhythmia requiring treatment, pulmonary hypertension, or chronic pulmonary disease requiring oxygen, venous thrombosis.
* Stroke or transient ischemic attack (TIA) in the 12 months before screening.
* Major depressive illness in the last 3 years; any history of severe psychiatric illness (eg, schizophrenia).
* Multiple sclerosis or any other demyelinating disease.
* Any of the following laboratory abnormalities:

  * Hemoglobin <8.5 g/dl (international system units [SI]: <85 g/L).
  * Neutrophils <1500/mm3 (SI: < 1.5 x 109/L).
  * White blood cell (WBC) count <3,000/mm3 (SI: < 3.0 x 109/L).
  * Platelets <80,000 mm3 (SI: 80 x 109/L).
  * International normalized ratio (INR) >1.5.
  * Serum creatinine >1.5 x the upper limit of normal.
* Has a current bacterial, parasitic, fungal, viral, or mycobacterial infection, or any major episode of infection requiring hospitalization or treatment with intravenous (IV) antibiotics within 4 weeks prior to the screening visit, and/or oral antibiotics within 2 weeks prior to screening visit and at any time during the screening period.
* Serological evidence of human immunodeficiency virus (HIV), hepatitis B surface antigen (HbsAg), or hepatitis C (HCVAb) at Screening (note: HCV subjects with undetectable viral load will be eligible).
* Clinically significant findings on 12-lead ECG such as, but not limited to, 2nd or 3rd degree AV block, prolongation of QRS complex over 120 msec, or QTcF interval ≥450 msec for males and ≥470 msec for females.

Medications of exclusion:

* Non-steroidal anti-inflammatory drugs (NSAIDs) daily.
* Subjects on anti-coagulation therapy within 28 days prior to screening and through Day 56.

Note: (A daily dose of ASA 81mg, taken for cardio prophylaxis, is considered acceptable to be continued during the study.)

* Topical (i.e., enema or suppository) mesalamine or steroid within 14 days prior to screening endoscopy.
* Azathioprine, 6-mercaptopurine, or methotrexate within the 28 days prior to screening.
* Any prior use of mycohphenolic acid, tacrolimus, sirolimus, cyclosporine, thalidomide
* Any prior use of biologics: rituximab, efalizumab, anti-integrines (natalizumab, vedolizumab, etrolizumab), TNF antagonists (infliximab, , golimumab, certolizumab pegol), anti-IL-12/23 (ustekinumab, guselkumab, risankizumab, or mirikizumab) ≤ 3 months prior to first dosing or ≤ 5 elimination half-lives prior to first dosing (whichever is shorter).
* Any prior use of small molecules: JAK inhibitors (tofacitinib, baricitinib, upadacitinib, or other) or S1P receptor modulator (fingolimod, ozanimod, etrasimod) ≤ 3 months prior to first dosing or ≤ 5 elimination half-lives prior to first dosing (whichever is shorter).
* Use of PPI (proton pump inhibitor) during the study (Should be discontinued 72 hours prior to Day 1).
* Use of prescription medications started or with a dose adjustment within 4 weeks prior to study screening, or over-the-counter medications or supplements started or with a dose adjustment within 2 weeks prior to study screening. Medications under Inclusion Criterion #5 are not included. Short-term administration of drugs for acute conditions are acceptable.
* Anti-diarrheal medications are not allowed within 48 hours of screening and throughout the study.
* Participated in another clinical trial of an investigational drug (or medical device) within 30 days prior to screening or is currently participating in another trial of an investigational drug (or medical device).
* Subjects with planned hospitalization or surgery during the study.
* Subject has known sensitivity to any of the products or components to be administered during dosing.
* Has previously received PL8177.
* History of alcohol or drug abuse and/or positive drug test at screening (with exception of marijuana if legal within the state and no drug abuse is noted in the PI's assessment)
* Positive TB or COVID 19 test. Note: Patients with positive TB results who had active or latent TB in the two years preceding the screening visit and who were treated for TB can participate in study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of PL8177 compared to placebo in patients with active UC. | Baseline through Study Completion (Week 12).
  Adverse events (AEs) will be collected from the time of signing the informed consent form (ICF). All subjects who are randomized will be monitored for AEs until the time they leave the study.
To compare the proportion of subjects achieving Mayo Endoscopic Subscore of ≤ 1 point (0 or 1) between PL8177 and placebo after 8 weeks of treatment. | Time Frame: Mayo Endoscopic Subscore will be evaluated at Week 8.
  Efficacy will be determined through the use of the Mayo Endoscopic Subscore.

OTHER OUTCOMES:
Summarize and evaluate the efficacy of PL8177 compared to placebo on histologic-endoscopic mucosal improvement | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo on histologic-endoscopic mucosal improvement (HEMI) after 8 weeks of treatment. Histologic-Endoscopic Mucosal Improvement is defined as MES of ≤ 1 point and a Geboes score ≤ 3.1.
Summarize and evaluate the efficacy of PL8177 compared to placebo on endoscopic remission | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo on endoscopic remission defined as MES = 0
Summarize and evaluate the efficacy of PL8177 compared to placebo on histologic remission | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo on histologic remission after 8 weeks of treatment (Geboes score ≤ 3.1)
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the Ulcerative Colitis Endoscopic Index of Severity | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the Ulcerative Colitis Endoscopic Index of Severity (UCEIS) after 8 weeks of treatment.
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the change in sum scores of segmental endoscopic disease severity for both the segmental MES and segmental UCEIS | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the change in sum scores of segmental endoscopic disease severity for both the segmental MES and segmental UCEIS (rectum, sigmoid colon, descending colon) from baseline to Week 8.
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the fecal calprotectin levels | Baseline through Week 8 (Day 57)
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the fecal calprotectin levels between baseline and Day 56/Week 8
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the Stool Frequency Subscore | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the Stool Frequency Subscore (SFS) after 8 weeks of treatment
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the Rectal Bleeding Subscore | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the Rectal Bleeding Subscore (RBS) after 8 weeks of treatment
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the 32-item Inflammatory Bowel Disease Questionnaire | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the 32-item Inflammatory Bowel Disease Questionnaire (IBDQ- 32) questionnaire after 8 weeks of treatment
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the Patient Reported Outcome | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the Patient Reported Outcome (PRO-2) after 8 weeks of treatment.
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the proportion of patients that have a clinical response | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the proportion of patients that have a clinical response defined as a reduction from baseline in the 3-component Mayo score of ≥ 2 points and ≥ 30% reduction from baseline with an accompanying decrease in RBS of ≥ 1 point or absolute RBS of ≤ 1 point.
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the proportion of patients that achieve clinical remission | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the proportion of patients that achieve clinical remission defined as a 3-component Mayo score of ≤ 2 with SFS = 0 or 1; RBS = 0; Centrally read endoscopy subscore = 0 or 1 (score of 1 modified to exclude friability) after 8 weeks of treatment.
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the intra-subject change in rectosigmoid disease | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the intra-subject change in rectosigmoid disease (per the MES) after 8 weeks of treatment
Summarize and evaluate the efficacy of PL8177 compared to placebo based on the overall global improvement | Baseline through Week 8
  Summarize and evaluate the efficacy of PL8177 compared to placebo based on the overall global improvement across efficacy parameters, summing the number of efficacy endpoints that improved

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jordan, VP Clinical Operations, Study Director — Telephone: 609-598-1786; Email: rjordan@palatin.com
Locations (14):
- United States (14):
  - Del Sol Research Management, LLC, Tucson, Arizona
  - Gastro Care Institute, Lancaster, California
  - Valiance Clinical Research, Tarzana, California
  - Advanced Research LLC, Coral Springs, Florida
  - IHS Health Research/Gastro Health, Kissimmee, Florida
  - Orlando Health, Inc., Orlando, Florida
  - Kansas Gastroenterology, Wichita, Kansas
  - Gastroenterology Clinic of Acadiana, Lafayette, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Allied Health Clinical Research Organization, LLC - Englewood, Englewood, New Jersey
  - Allied Digestive Health LLC, Freehold, New Jersey
  - Allied Health Clinical Research Organization, LLC, Jackson, New Jersey
  - Weill Cornell Medicine - Jill Roberts Center for Inflammatory Bowel Disease, New York, New York
  - UPMC Presbyterian, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No